

# Protocol for non-interventional studies based on existing data

| Document Number: | c30699487-01 |
|---|---|
| BI Study No.: | 1237-0094 |
| BI Investigational Product(s): | Tiotropium bromide + Olodaterol |
| Title: | Effectiveness and Safety of Maintenance Treatment with Combination of Tiotropium and Olodaterol in comparison to Maintenance Treatment with a Combination of Inhaled Corticosteroids, Long-acting β2 Agonists and Long-acting Muscarinic Antagonists in COPD Patients |
| Title for lay people: | Comparative Effectiveness and Safety of Tiotropium and Olodaterol in comparison to Triple Therapy |
| Date of last version of protocol: | NA |
| EU PAS Register No: | Not applicable |
| Marketing authorization holder(s): | |
| Author/Responsible<br>Parties/BI contact<br>person: | Authors/Responsible parties: |
| | Tel.:<br>Mobil:<br>Fax:<br>Email: |
| Country(-ies) of study: | United States |
| Status: | Protocol Final Version 1 |

## **Boehringer Ingelheim**

Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

c30699487-01


| EU-QPPV: only applicable for PASS | Not applicable | |
|---|---|---|
| Signature of EU-QPPV: only applicable for PASS | Not applicable | |
| Version: 1.0 | | Date : 12 Dec 2019 |
| | Page 1 | of 57 |
| | | ential information e or more of its affiliated companies. All rights reserved. ed, published or otherwise used without prior written permission |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ABSTRACT**

| Name of company: Boehringer Ingelheim Name of product: Spiole Name of active ingredie Tiotropium bromide + | nt: | | Boehringer<br>Ingelheim |
|---|---|---|---|
| D ( 11 ) | | W . W | W |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 December 2019 | 1237-0094 | 1.0 | NA |
| | heim International GmbH | confidential information I or one or more of its affiliated compreproduced, published or otherwise used with | |
| Title of study: | Title of study: Effectiveness and Safety of Maintenance Treatment with Combination of Tiotropium and Olodaterol in comparison to Maintenance Treatment with a Combination of Inhaled Corticosteroids, Long-acting β2 Agonists and Long acting Muscarinic Antagonists in COPD Patients | | |
| Team member<br>Epidemiology: | | | |
| Project team: | (P | Principal Investigator) | |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of company: Boehringer Ingelhei Name of product: Sp Name of active ingree Tiotropium bromide | iolto<br>dient: | | Boehringer Ingelheim |
|---|---|---|---|
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 December 2019 | 1237-0094 | 1.0 | NA |

#### Proprietary confidential information

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

# Rationale and background:

The treatment of COPD involves multiple therapies, including long-acting β2 agonists (LABA) (with and without inhaled corticosteroids (ICS) and long-acting muscarinic antagonists (LAMA), with combinations of these drugs now formulated into single inhalers.

There are recommendations to restrict triple therapy use further, to only patients who are likely to respond to ICS (such as those with asthma-COPD overlap or patients with high risk of exacerbations and elevated blood eosinophils [P15-08642, P07-11503, R19-3048]. There is an increasing body of evidence suggesting that ICS are particularly effective at reducing the incidence of COPD exacerbations in patients only with a very high blood eosinophil concentration, but not in normal levels [P18-09975]. Hence there is a clear need for better evidence on specific patient populations upon which to base treatment recommendations.

This non-interventional study aims to assess the comparative effectiveness of combination Tiotropium and Olodaterol (Tio+Olo) (FDC) compared to combination LAMA/LABA and ICS (fixed or open), and to explore whether this varies across COPD sub populations defined by exacerbation risk. The intended audiences are payers and prescribers. The results from the study will be published in the scientific literature.

| Name of company: | | | Boehringer<br>Ingelheim |
|---|---|---|---|
| Boehringer Ingelheim | | | VIIIIIV Ingelheim |
| Name of product: Spiol | Name of product: Spiolto | | |
| Name of active ingredic | ent: | | |
| Tiotropium bromide + | Olodaterol | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 December 2019 | 1237-0094 | 1.0 | NA |
| © 2019 Boehringer Inge<br>This document may not - i | lheim International GmbH | confidential information I or one or more of its affiliated compreproduced, published or otherwise used with | panies. All rights reserved. |
| objectives: | In the primary objective is to compare the effectiveness of maintenance theraps initiation with the combination treatment Tiotropium and Olodaterol (Tio+Olo) compared with any LABA/LAMA/ICS combination in COPD and time to community acquired pneumonia. The primary objective is to assess the association between maintenance therapy initiation with the combination in COPD and time to community acquired pneumonia. Additionally, we will assess differences between Tio+Olo vs any LABA/LAMA/ICS in healthcare utilization and all-cause and COPD-specific cost overall and by care settings. | | |
| Study design: | | cohort design will be used, with and reweighting of time-condition | |

| Name of company: | | | Boehringer |
|---|---|---|---|
| Boehringer Ingelheim | | | Ingelheim |
| Name of product: Spiolto | | | |
| Name of active ingredie | ent: | | |
| Tiotropium bromide + | | | |
| Troughtum Gromae | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 December 2019 | 1237-0094 | 1.0 | NA |
| | lheim International GmbH | confidential information I or one or more of its affiliated compreproduced, published or otherwise used with | |
| | who received Tio+Ol January 2013 until 31 time of cohort extract and decrease the likel will only include patiexclude all patients windex date or lung car any time prior to the Patients will have at I cohort entry date to a of baseline covariates treatment, other changend of the individual' whichever occurs firs following the index d Additional restriction showing eosinophil let | The cohort will consist of all patients in the HIRD with a diagnosis of COPD who received Tio+Olo or combination LABA/LAMA/ICS treatment from 1 January 2013 until 31 March 2019 (or the most recent date available at the time of cohort extraction). To increase the likelihood of a diagnosis of COPD and decrease the likelihood of including misdiagnosed asthma patients, we will only include patients 40 years of age or older on the index date and exclude all patients with a diagnosis of asthma within the year prior to the index date or lung cancer, interstitial lung disease, or lung transplantation at any time prior to the index date. Patients will have at least one year of medical history information prior to the cohort entry date to allow the identification of new use and the measurement of baseline covariates. Patients will be followed until switching to the other treatment, other changes in therapy, discontinuation of COPD treatment, the end of the individual's health plan eligibility, or the end of the study period, whichever occurs first. Main analyses will be limited to the first year following the index date. Additional restriction to individuals who have laboratory test result data | |
| Study data source: | The HealthCore Integ | grated Research Database <sup>SM</sup> (HII | RD) |
| Expected study size: | Overall: New users of Tio+Olo: 5,458 New users of LABA/LAMA/ICS: 42,361 With eosinophil result data: New users of Tio+Olo: 2,198 New users of LABA/LAMA/ICS: 15,712 | | |
| Main criteria for inclusion: | either as a fixed-dose<br>(LABA/ICS + LAMA<br>March 2019. | Do on the same date or of LABA, LAMA and ICS, combination (LABA/LAMA/ICS) or free combination (A, etc), on the same date between January 2013 and prior to first maintenance inhaler and age ≥ 40 years | |

# Boehringer Ingelheim

# Protocol for non-interventional studies based on existing data BI Study Number 1237-0094


c30699487-01

| Name of company: Boehringer Ingelheim Name of product: Spiole | to | | Boehringer Ingelheim |
|---|---|---|---|
| Name of active ingredie | nt: | | |
| Tiotropium bromide + Olodaterol | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 December 2019 | 1237-0094 | 1.0 | NA |
| | heim International GmbH | confidential information<br>I or one or more of its affiliated compreproduced, published or otherwise used with | |
| Main criteria for exclusion: | -Less than one year of medical history information prior to the date of combined treatment initiation (index date) -Lung cancer, interstitial lung disease, or lung transplantation at any time prior to the index date | | |
| | -Asthma diagnosis within one year prior to the index date | | |
| Comparison groups: | Initiating Tio+Olo compared to initiating LABA/LAMA/ICS therapy | | |
| Expected duration of exposure: | Analyses will be limited to one year following the index date for the primary and secondary analyses. Sensitivity analyses will use all available exposure data. | | |

## TABLE OF CONTENTS

| TITLE I | PAGE | 1 |
|---|---|---|
| ABSTRA | ACT | 3 |
| TABLE | OF CONTENTS | 8 |
| 1. | LIST OF ABBREVIATIONS AND TERMS | 10 |
| 2. | RESPONSIBLE PARTIES | 12 |
| 3. | AMENDMENTS AND UPDATES | |
| 4. | MILESTONES | 12 |
| 5. | RATIONALE AND BACKGROUND | |
| 6. | RESEARCH QUESTIONS AND OBJECTIVES | |
| 7. | RESEARCH METHODS | |
| 7.1 | STUDY DESIGN | |
| 7.2 | SETTING | |
| 7.3 | SUBJECTS | |
| 7.4 | VARIABLES | |
| 7.4.1 | Exposures | |
| 7.4.2 | Outcome(s) | |
| 7.4.2.1 | Primary outcome(S) | |
| 7.4.2.2 | Secondary outcome(s) | |
| 7.4.3 | Covariates | 17 |
| 7.5 | DATA SOURCES | |
| 7.6 | BIAS | |
| 7.7 | STUDY SIZE | |
| 7.8 | DATA MANAGEMENT | |
| 7 <b>.</b> 9 | DATA ANALYSIS | |
| 7.9.1 | Main analysis | |
| 7.10 | QUALITY CONTROL | 24 |
| 7.11 | LIMITATIONS OF THE RESEARCH METHODS | |
| 7.12 | OTHER ASPECTS | |
| 8. | PROTECTION OF HUMAN SUBJECTS | <b>2</b> 6 |
| 9. | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 27 |
| 10. | PLANS FOR DISSEMINATION AND COMMUNICATION OF STUDY RESULTS | Z |
| 11. | REFERENCES | |
| 11.1 | PUBLISHED REFERENCES | |
| 11.1<br>11.2 | UNPUBLISHED REFERENCES | |
| 1 1 . Z | UNI UDIJABINI REPERENUEN | |

| Boehringer Ingelheim | |
|---------------------------------------------|---------------------|
| Protocol for non-interventional studies bas | ed on existing data |
| BI Study Number 1237-0094 | |


c30699487-01

| 12. | FUNDING | 33 |
|---------|----------------------------------------|----|
| | ANNEX | |
| | : LIST OF STAND-ALONE DOCUMENTS | |
| | : ENCEPP CHECKLIST FOR STUDY PROTOCOLS | |
| | :ADDITIONAL INFORMATION | |
| | 3.1: DEFINITION OF STUDY EXPOSURES | |
| ANNEX 3 | 3.2: DEFINITIONS OF STUDY OUTCOMES | 42 |
| | 3.3: DEFINITIONS OF STUDY COVARIATES | |
| ANNEX 3 | 3.4:STATISTICAL CONSIDERATIONS | 57 |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. LIST OF ABBREVIATIONS AND TERMS

AE Adverse Event

BI Boehringer Ingelheim

BMI Body Mass Index

CI Confidence Interval

COPD Chronic obstructive pulmonary disease

CPRD Clinical Practice Research Datalink

DSAs Data Sharing Agreements

ED Emergency Department

EMA European Medicines Agency

FDC Fixed Dose Combination

GVP Guideline on Good Pharmacovigilance Practices

HIPAA Health Insurance Portability and Accountability Act

HIRD HealthCore Integrated Research Database

ICD-10 International Classification of Disease, Version 10

ICS Inhaled corticosteroids

IR Incidence Rate

IRB Institutional Review Board

ITT Intention to treat

LABA Long-acting beta2-agonist

LAMA Long-acting muscarinic antagonists

N Number

PHI Protected Health Information

PS Propensity score

PSTAT Project Statistician

PY Person-years at risk

RR Rate Ratio

TIO+OLO Tiotropium+Olodaterol

# Boehringer Ingelheim Protocol for non-intervention

# Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

 c30699487-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TM Epi Team Member Epidemiology

 $cells/\mu L \qquad \qquad Microliter$ 

US United States

UTS Up-to-standard

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. RESPONSIBLE PARTIES

(Principal Investigator)

Tel:

### 3. AMENDMENTS AND UPDATES

There are currently no amendments to the protocol.

### 4. MILESTONES

| Milestone | Planned date |
|---|---|
| Start of data collection: | August 1, 2019 |
| Data extraction and coding | |
| End of data collection: | Not applicable. This study is an observational study based on existing data. |
| Study progress report(s) as referred in Article 107 m(5) of Directive 2001/83/EC: | Not applicable |
| Interim report(s) of study results: | Not applicable |
| Registration in the EU PAS register | Not applicable |
| Final report of study results: | April 2020 (Preliminary results: 19 December 2019) |

BI Study Number 1237-0094

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. RATIONALE AND BACKGROUND

The treatment of COPD involves multiple therapies, including Long-acting  $\beta$ 2 agonists (LABA) (with and without inhaled corticosteroids (ICS) and long-acting muscarinic antagonists (LAMA), with combinations of these drugs now formulated into single inhalers.

Several trials compared a single-inhaler triple therapy with an ICS/LABA and a LAMA respectively and found greater benefit with triple FDC [P19-08111]. However, they represent a limited view of the patients who could potentially use these treatments so that a real-world study of patients who are representative of clinical practice is of interest.

There are recommendations to restrict triple therapy use further, to only patients who are likely to respond to ICS (such as those with asthma-COPD overlap or elevated blood eosinophils [P15-08642). There is an increasing body of evidence suggesting that ICS are particularly effective at reducing the incidence of COPD exacerbations in patients only with a very high blood eosinophil concentration, but not in normal levels [P18-09975]. Hence there is a clear need for better evidence on specific patient populations upon which to base treatment recommendations.

This non-interventional study aims to assess the comparative effectiveness of combination Tiotropium and Olodaterol (Tio+Olo) (FDC) compared to combination LAMA/LABA and ICS (fixed or open) This study will provide useful data on the relative benefits of different combinations in treating COPD patients The intended audiences are payers and prescribers. The results from the study will be published in the scientific literature.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. RESEARCH QUESTIONS AND OBJECTIVES

The goal of this study is to investigate the risk of COPD exacerbations, community acquired pneumonia, and health care utilization in patients treated with Tio+Olo in comparison to patients treated with ICS/LABA/LAMA. All analyses will be conducted for the total population, as well as in sub-groups of patients under (1) high- or low risk of exacerbation based on previous history of exacerbations in the year preceding cohort entry (cut-off: 0-1 vs 2+ exacerbations [P07-11503], (2) circulating eosinophils (cut-off B-Eos 300 cells/uL, [P18-09975]), and (3) as an exploratory analysis, a combination of exacerbation history and circulating eosinophils.

#### **Primary objectives:**

The primary objective is to compare the effectiveness of new use of maintenance therapy initiation with the combination treatment Tiotropium and Olodaterol (Tio+Olo) compared with new use of LABA/LAMA/ICS combination in COPD as the time to the first COPD exacerbation.

#### Secondary objective:

The secondary objective is to assess the association between maintenance therapy initiation with the combination treatment (Tio+Olo vs any LABA/LAMA/ICS combination in COPD and time to community acquired pneumonia.

#### **Exploratory objective:**

To assess differences between Tio+Olo vs any LABA/LAMA/ICS in all-cause and COPD-specific healthcare utilization and cost overall and by care setting.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RESEARCH METHODS

#### 7.1 STUDY DESIGN

Population-based incident new-user cohort design.

#### 7.2 SETTING

The study will be conducted using administrative healthcare claims and laboratory result data captured in the HealthCore Integrated Research Database (HIRD; details in Section 7.5). The observation period will be from January 2013 until the most recent date available at the time that the cohort is extracted (estimated March 2019).

#### 7.3 SUBJECTS

The study cohort will be formed based on the following entry criteria.

#### **Inclusion Criteria:**

- 1. At least one prescription for Tio+Olo or a LABA/LAMA/ICS combination between 1 January 2013 and 31 March 2019.
  - a. For Tio+Olo users, the first dispensing of Tio+Olo will be defined as the index date.
  - b. LABA/LAMA/ICS use can occur either in free or fixed combinations. The first date when all three medications are used based on either concurrent or overlapping dispensings in the pharmacy claims data will be defined as the index date.
- 2. At least one diagnosis of COPD at any time prior to the index date.
- 3. At least one year of continuous medical and pharmacy health plan eligibility prior to the index date will be required to allow a baseline period for the covariates and identification of new use of the study drugs.

#### **Exclusion Criteria:**

- 1. To increase the likelihood of a true diagnosis of COPD, we will exclude:
  - a. All patients less than 40 years of age on the index date, and
  - b. All patients with a diagnosis of asthma in the year prior to the index date
- 2. To limit the population to those without severe lung compromise outside of COPD, we will exclude individuals with lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date
- 3. To restrict the cohort to new users of Tio+Olo or LABA/ICS, we will exclude any individual with use of either Tio+Olo, LABA/ICS, or LABA/LAMA/ICS combination therapy in free or fixed form for at least one year prior to the index date.

Outpatient laboratory data is available for a subset of patients. Some analyses will be further restricted to the subset of the population with at least one laboratory result showing circulating eosinophil levels within six months before the index date.

Individuals in the study cohort will be followed from the index date until the earliest of the date of a switch in treatment, addition of ICS for the Tio+Olo group, discontinuation of

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

COPD treatment, the end of the study period, or the end of continuous health plan eligibility. Main analyses will be further limited to the first year after cohort entry, with sensitivity analyses considering all available data.

#### 7.4 VARIABLES

#### 7.4.1 Exposures

The exposure measures are based on pharmacy dispensings of the study medications, namely Tio+Olo and LABA/LAMA/ICS combination therapy. As described in the data analysis section, the as-treated analysis, which is the main analysis, will consider continuing exposure of the initial treatment of Tio+Olo or LABA/LAMA/ICS within the treated groups defined by the days supply recorded at the time of pharmacy dispensing, allowing for a gap between dispensings of up to 15 days. This gap is allowed in consideration of plausible delays in obtaining medication refills and continued use beyond the days supplied where medication has been missed due to imperfect adherence, and will be varied in sensitivity analyses (see Section 7.9.2). Codes used to identify study medications are included in Annex 3.1.

The treatment segment ends at the earliest of the following events:

- 1. Fifteen days after the end of the observed days supply for the medication received on the index date without a subsequent dispensing of COPD medication (i.e., discontinuation)
- 2. Initiation of triple therapy (i.e., addition of ICS to Tio+Olo or a LAMA to LABA/ICS (i.e., treatment escalation, applies to Tio+Olo only)
- 3. Any other change in use of study medication by active ingredient, inclusive of a change to a different combination therapy, change from a fixed form to a free form combination therapy, or a change from combination therapy to monotherapy (i.e., switch)

Changes in dose for medications started on the index date will not impact the end of the treatment segment. Codes used to identify study medications are included in Annex 3.1.

#### **7.4.2 Outcome(s)**

#### 7.4.2.1 Primary outcome(S)

The primary outcome event for effectiveness is the first COPD exacerbation to occur after cohort entry. The event is defined as follows:

- Severe exacerbation:
  - o Hospitalization with a principal discharge diagnosis of COPD.
- Moderate exacerbation:
  - o An ED visit with a discharge diagnosis of COPD and/or
  - o Dispensing of an antibiotic and an oral corticosteroid on the same day

Time to the first COPD exacerbation will be measured from cohort entry until the occurrence of a hospitalization for COPD (severe exacerbation) or ED visit for COPD with the prescription of an antibiotic and/or an oral corticosteroid on the same day (moderate exacerbation). Severe and moderate exacerbations will be considered as a composite for main analyses. Sensitivity analyses will stratify by exacerbation severity.

Although there is precedent for defining moderate exacerbation based on use of antibiotics for a respiratory infection without requiring concomitant oral corticosteroids, we have chosen

a more restrictive definition of exacerbation. Because diagnoses listed on outpatient claims often correspond to a patient's past medical history in addition to acute problems, we expect limited ability to capture the indication for which antibiotics are prescribed. As such, including antibiotics alone as a case definition for exacerbation would introduce potentially substantial misclassification of outcome where antibiotics were truly given for non-respiratory infections. Given that our analyses will yield estimates on a ratio measure, non-differentially reduced sensitivity is a less important threat to validity than reduction of outcome specificity, which produces an expectation of bias towards the null hypothesis. In order to test our assumptions that the sensitivity of our outcome definition is not differential between the Tio+Olo and LABA/ICS groups, we would produce counts of patients with antibiotics alone during follow-up, and determine whether the proportion of potential exacerbations that we excluded through this design decision is comparable across groups.

#### 7.4.2.2 Secondary outcome(s)

The secondary outcome is the occurrence of the first hospitalization for community-acquired pneumonia (serious pneumonia). Pneumonia will be defined using ICD-9-CM diagnoses 481.x-486.x; 487.0, 507.x, 507.0, 507.1, 507.8, 510.0, 510.9, 511.0, 513.0, 514.x, 517.1, 519.8, 530.84, and ICD-10 diagnosis codes J10.0; J11.0; J12-J18; J22; J69; J85.0; J85.1; J86. This definition has been used successfully in COPD [P07-09514; P16-10095].

#### 7.4.3 Covariates

Patient characteristics at baseline will be assessed for Tio+Olo and LABA/LAMA/ICS user overall and stratified by history of exacerbation, circulating eosinophils, subgroups defined by both exacerbation and eosinophil levels.

We will identify and describe the following demographic characteristics as of the index date:

- Sex
- Age (years, as both a categorical and a continuous variable)
- Calendar year of cohort entry

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Season of index date (winter, spring, summer, fall)
- US census region of residence
- Insurance type (e.g., Commercial, Medicare)

Additional characteristics will be defined during the 12-month pre-index baseline period:

- Number of previous COPD treatments
- Specific previous COPD treatments
  - o LAMA monotherapy
  - o LABA monotherapy
  - o ICS monotherapy
  - o LAMA/ICS combination therapy
  - o LABA/ICS combination therapy
- Previous acute COPD exacerbation (measured both overall and in the 30 days prior to cohort entry), categorized as 0, 1, or 2+.
  - All exacerbations (Moderate+Severe)
  - o ED visits or dispensings of inhaled corticosteroids/antibiotics (Moderate)
  - o Hospitalizations (Severe)
- Use of other respiratory drugs in the 12-month pre-index period:
  - o Short-acting beta-agonists
  - o Anticholinergics
  - o Methylxanthines
  - o Muscarinic antagonists
  - o Short-acting muscarinic antagonists
- Use of antibiotics for a respiratory condition (e.g., azithromycin)

Chronic comorbidities will be defined using diagnoses identified during all available data prior to the index date, and will include:

- Cardiovascular disease
- Charlson comorbidity index
- Diabetes
- Thyroid disease
- Renal failure
- Autoimmune disease
- Pneumonia
- Obesity\*
- Alcohol use disorder\*
- Tobacco use or cessation counselling\*
- Cancer (excluding basal cell carcinoma)
- \* We anticipate limited capture of lifestyle variables known to be risk factors and potential confounders, including obesity, smoking status and excessive alcohol consumption. Although we will describe them as identified in the HIRD, bias analyses to examine the extent to which residual confounding may impact results are also planned.

Additionally to the covariates defined above, we will use the high-dimensional approach to identify variables entering a time-conditional propensity score.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Sub-populations will include patients with high or low circulating eosinophils (B-Eos 300 cells/uL [P18-09975] as identified based on the laboratory result value that is closest but prior to the index date (within 6 months). Additional stratification will include previous history of exacerbations in the year preceding cohort entry (with exacerbation history defined as either 1 + hospitalization or 2 + exacerbations in emergency department or outpatients settings), and among those without a history of exacerbation at baseline, based on circulating eosinophil results as noted above. However, number of patients with baseline exacerbations and data available on B-Eos is very low (see section 7.7) and therefore analysis would not be meaningful and will not be performed.

#### 7.5 DATA SOURCES

This study will be conducted using the HIRD, a large administrative healthcare database maintained by HealthCore for use in health outcomes and pharmacoepidemiologic research. The HIRD includes longitudinal medical and pharmacy claims data from health plan members across the United States (US). Member enrolment, medical care (professional and facility claims), outpatient prescription drug use, outpatient laboratory test result data, and health care utilization may be tracked for health plan members in the database dating back to January 2006, and with diagnoses recorded in International Classification of Disease, Version 10 (ICD-10) since October, 2015. Laboratory result data are additionally available for those tests that have been performed using two large, national reference laboratories (Quest and LabCorp) [R14-4278]. The database has been used for the study of numerous diseases, including studies of COPD [R19-2324; R19-2321; R19-2323; R19-2322; P15-11025; P14-12233]

#### **7.6 BIAS**

Several potential biases are inherent to any observational study in the HIRD. In the absence of randomization, confounding by indication could be an issue. Controlling by propensity score should limit this bias, but can control only for measured covariates and may produce estimates that are impacted by residual confounding. This is of particular importance in the case of lifestyle factors that are less critical to insurance billing and thus poorly captured in claims data. Quantitative bias analyses can formally describe the extent to which these issues are present, but bias analysis parameters are informed by literature and clinical expert opinion. As such, the accuracy of bias corrected analyses is limited by the accuracy of the assumptions that inform them [R19-3031].

Second, there is the possibility of information bias due to misclassification of the outcomes or exposure or missing data, especially, differential missingness of some data (e.g. eosinophils, which may only be measured in sicker patients). The prescriptions dispensed by a pharmacy but not taken by patients could lead to misclassification of exposure. Pharmacy dispensing data does bring us one step closer to patient use than physician prescribing given that the patient has taken the effort to obtain the medication as instructed, however, information such as indication can only be inferred based on diagnostic patterns.

#### 7.7 STUDY SIZE

Preliminary patient counts in the HIRD are shown here:

| | Tio+Olo | | ICS/LAB | A/LAMA |
|---------------------------------|---------|-------|---------|--------|
| | N | % | N | % |
| New users | 8,233 | 100.0 | 82,534 | 100.0 |
| At least 12 months of | | | | |
| pre-index eligibility | 6,263 | 76.1 | 50,153 | 60.8 |
| Age 40 + | 6,126 | 97.8 | 48,267 | 96.2 |
| At least 1 diagnosis of COPD | 5,469 | 89.3 | 42,227 | 87.5 |
| At least 1 eosinophil % result | • | | | |
| prior to the index date | 2,207 | 40.4 | 15,699 | 37.2 |
| Eosinophil result (N, % of | | | | |
| those with a result) | | | | |
| 0-2% | 1,059 | 48.0 | 7,488 | 47.7 |
| 2-4% | 745 | 33.8 | 5,136 | 32.7 |
| 4%+ | 403 | 18.3 | 3,075 | 19.6 |
| Eosinophil result, patients | | | | |
| with low exacerbation | | | | |
| history(0 inpatient and 0-1 | | | | |
| outpatient events at baseline, | | | | |
| N, %) | | | | |
| <300 cells/uL | 1,381 | 30.0 | 9,516 | 27.3 |
| ≥300 cells/uL | 481 | 10.5 | 3,481 | 10.0 |
| Unknown | 2,739 | 59.5 | 21,813 | 62.7 |
| Eosinophil result, patients | | | | |
| with high exacerbation history | | | | |
| (1 + inpatient or 2 + outpatien | | | | |
| t events at baseline, N, %) | | | vents | |
| <300 cells/uL | 226 | 26.0 | 1,888 | 25.5 |
| ≥300 cells/uL | 105 | 12.1 | 707 | 9.5 |
| Unknown | 537 | 61.9 | 4,822 | 65.0 |

In a recent analysis of the risk of exacerbations based on Clinical Practice Research Datalink (CPRD), a total of 2,000 patients per cohort detected a 15% difference in risk of a first exacerbation (hazard ratio 0.85) with over 90% power. As such, overall analyses and analyses that are stratified based on the presence of claims-based indicators of exacerbation are expected to have adequate power. Analyses limited to individuals with specific eosinophils will be more limited. Given low expected sample size, stratification by eosinophil analysis within individuals with exacerbations at baseline will not be performed by Eosinophil categories.

BI Study Number 1237-0094

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.8 DATA MANAGEMENT

All statistical analysis for the study will be conducted using SAS version 9.4 or higher (SAS Institute, Cary, NC). All sensitive data pertaining to the study will be stored on secured servers with access only permitted by approved study team members.

A number of Information Security policies are enforced, audited, and in place at HealthCore, including complex password requirements and encryption systems. Security mechanisms and policies are in place HealthCore's facilities are standard corporate office space. Office space is segregated and managed by monitored electronic access. HealthCore areas which contain project and study-related documents are only access by HealthCore associates or contract personnel. All non-HealthCore associates must be accompanied by an associate at all times in order to enter these areas. All study related files are kept in locked cabinets and work areas. There are no visible labels or client listings viewable by any visitor or passerby. All passwords and user authentication mechanisms are forced changed at regular intervals and there is automatic locking of workstations after a short period of time (< 15 minutes).

Data Center space is permitted on an as required basis and monitored by electronic access. HealthCore maintains a cumulative record that indicates, for any point in time, the names of authorized personnel, their titles, and a description of their access privileges to the Data Center. Data access is restricted, monitored, logged, and audited. HealthCore's computer networks have been designed to separate patient or physician identified data from de-identified or masked data. Network security, firewalls, and password permissions control which HealthCore personnel have access to patient or physician identifiers. Unless the study protocol calls for patient or physician authorization or a waiver of authorization as granted by an IRB, no research analyst will have access to patient or physician identifiers within HealthCore's computer systems. All research analysis databases have been de-identified. HealthCore's Data Center is also physically secured by a controlled access facility, with only authorized personnel having access to network servers, tape libraries and other media that contains patient identifiers.

Research analysis files used by HealthCore do not contain patient or physician identifiers unless necessary to perform such research; if such is the case, access will be made after receipt of the patient's or physician's authorization or IRB waiver of such authorization has been granted. It is also HealthCore policy to provide for secure storage of study materials, including data, reports, and other files after the study is completed, with a destroy date assigned based on study requirements. HealthCore reviews data requirements for each study to assure that only the minimum of patient or physician information is obtained to answer the research question(s). For those studies where direct patient identifiers are needed for additional data collection such as medical chart abstracts, access to information will be limited to the greatest possible extent within the research team. Both structural and contractual safeguards reinforce policies to minimize the risk of breaching patient or physician privacy. The structural safeguards include a clearly defined data flow process. This process minimizes the risk of individual identifiers being improperly used or disclosed. The contractual safeguards include contractual binding to confidentiality of individuals involved in the research.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.9 DATA ANALYSIS

#### 7.9.1 Main analysis

All analyses will be presented for each group (Tio+Olo vs LABA/LAMA/ICS) overall and stratified as follows:

- History of exacerbation: 0 inpatient and 0-1 outpatient events
- History of exacerbation: 1 + inpatient or 2 + outpatient events
- Circulating eosinophils: B-Eos < 300 ug/mL
- Circulating eosinophils: B-Eos 300 ug/mL+
- History of exacerbation: 0 inpatient and 0-1 outpatient events & circulating eosinophils: B-Eos < 300 ug/mL
- History of exacerbation: 0 inpatient and 0-1 outpatient events & circulating eosinophils: B-Eos 300 ug/mL +

We will first describe formation of the study cohort. Patient characteristics at baseline in patients treated with Tio+Olo and patients treated with LABA/LAMA/ICS will be described using standard descriptive statistics. Because eosinophil levels may vary based on exacerbation, we will also provide a count and percentage of the number of individuals whose eosinophil results were recorded within 30 days of an exacerbation event.

High-dimensional propensity scores including both pre-specified and data-derived variables will then be calculated. We will use fine stratification and reweighting of the exposure propensity score to control for measured covariates [R19-3030]. Balance of patient characteristics between the cohorts will be described before and after propensity score application and compared using standardized differences (in the crude population and the reweighted pseudo-population). Standardized differences greater than 0.10 (10%) will be taken to indicate imbalance and further refinement approaches will be applied.

For the analysis of the primary objective, a Cox proportional hazard regression model will be used to perform an as-treated analysis that assesses the effect of current use of LABA-LAMA-ICS combination versus the Tio+Olo combination on the risk of a first COPD exacerbation. It will provide an estimate of the hazard ratio (HR) of a COPD exacerbation associated with LABA-LAMA-ICS use relative to Tio+Olo use, along with 95% confidence intervals (CI). Current use will be defined based on the days supply during the period of overlap, allowing a grace period of 15 days following the end of days supply to account for intermittent use. This approach allows consideration of exposure as time-dependent, accounting for the changes in exposure during the follow-up. In particular, this analysis excludes patients stopping one or more of the drugs prior to the index date.

Stratified analyses will use the same approach. Because not all individuals will have available laboratory result data available, fine stratification and reweighting by propensity score will be repeated within the subset of the cohort with available results to create weighted populations suitable for these stratified analyses. Potential effect-modification by B-Eosinophils and/or exacerbation history will be studied by comparing models with and without interaction terms and through qualitative consideration of differences in stratum-specific estimates.

#### Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

**** 

c30699487-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The analysis of the risk of pneumonia will also use a time-dependent Cox proportional hazard regression model with an as-treated approach, similar to that of the primary analysis.

In addition, we will repeat the primary effectiveness analysis on the time to exacerbation separately for moderate and severe exacerbations.

In terms of healthcare utilization, we will present continuous and categorical variables using standard descriptive statistics to describe total visits and total costs related to inpatient, outpatient, office visit, and emergency care as well as total pharmacy dispensings, distinct medications used, and pharmacy costs. Utilization and costs will be stratified to facilitate comparison between Tio+Olo and LABA/ICS, and presented by individual setting and as a composite. All-cause and COPD-specific data will be shown.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.10 **OUALITY CONTROL**

HealthCore operates observational research studies with the goal that the services provided to our clients are of high quality. To support this imperative we believe it is critical 1) to have dedicated training and quality resources and 2) that all talking points and major processes to be implemented with the study be approved by Boehringer Ingelheim in advance.

HealthCore's quality control program is centralized within the Regulatory Compliance Office. The Regulatory Compliance Office Manager is responsible for quality control and reports directly to the Vice President of Operations of HealthCore on all quality matters. HealthCore's quality system is organized around the Quality Manual, the quality checks within the project life cycle, and Standard Operating Procedures (SOPs). HealthCore has procedures for retention of protected health information (PHI) and project data. The study will be tracked at various levels to help ensure that all aspects including project delivery, infrastructure, quality processes, resource management, and financial issues are addressed. To help ensure the highest level of quality on every project, HealthCore has established several layers of quality assurance throughout the project lifecycle.

Role Based Control Checks: Each member of the team is responsible to perform thorough quality control checks on their work. In addition, the PI and Research Project Manager are also accountable for quality of all deliverables.

Quality Check Points: Centralized "checkpoints" have been implemented during the data management cycle to help ensure accurate translation of programming requests.

Quality Assurance Standards: Standard review procedures have been developed and are applied throughout the project lifecycle.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Automation: HealthCore has developed standard definitions of many variables and disease states and developed programs to apply these standards as needed on projects. These standards help ensure consistency, repeatability and accuracy for each project.

#### 7.11 LIMITATIONS OF THE RESEARCH METHODS

Several potential biases are inherent to any observational study in the HIRD. In the absence of randomization, confounding by indication could be an issue. Controlling for propensity to add the second treatment should limit this bias, but can control only for measured covariates and may produce estimates that are impacted by residual confounding. This is of particular importance in the case of lifestyle factors that are less critical to insurance billing and thus poorly captured in claims data. Quantitative bias analyses can formally describe the extent to which these issues are present, but bias analysis parameters are informed by literature and clinical expert opinion. As such, the accuracy of bias corrected analyses is limited by the accuracy of the assumptions that inform them.

Second, there is the possibility of information bias due to misclassification of the outcomes or exposure or missing data, especially, differential missingness of some data (e.g. eosinophils, which may only be measured in sicker patients). The prescriptions dispensed by a pharmacy but not taken by patients could lead to misclassification of exposure. Pharmacy dispensing data does bring us one step closer to patient use than physician prescribing given that the patient has taken the effort to obtain the medication as instructed, however, information such as indication can only be inferred based on diagnostic patterns.

#### 7.12 OTHER ASPECTS

None

BI Study Number 1237-0094

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. PROTECTION OF HUMAN SUBJECTS

HealthCore maintains Data Sharing Agreements (DSAs) and Business Associate Agreements with covered entities that provide protected health information (PHI) incorporated into the HealthCore Integrated Research Database (HIRD). HealthCore's access, use, and disclosure of PHI are in compliance with the Health Insurance Portability and Accountability Act (HIPAA) Privacy Rule [45 CFR Part 160 and Subparts A and E of Part 164]. HealthCore does not access, use, or disclose PHI other than as permitted by HIPAA and its Business Associate Agreements. When using PHI for research, this typically means we will use PHI to create limited data sets for research, or when that is not feasible we may obtain a specific waiver of the HIPAA authorization requirements from an Institutional Review Board (IRB). HealthCore also takes into consideration other federal and state laws and regulations that might limit use of certain types of data more than HIPAA, including those laws related to identifiable records related to substance abuse and human immunodeficiency virus.

The current study is designed as an analysis based on medical and pharmacy claims data from a large insured population in the United States (US). There is no active enrollment or active follow-up of study subjects, and no data will be collected directly from individuals.

At no time during the conduct of this study will HealthCore provide patient or provider identifying information to Boehringer Ingelheim All data and/or results will be in an aggregated and de-identified format. Data variables with values  $\leq 10$  will be reported only as " $\leq 10$ ." Boehringer Ingelheim will not attempt to re-identify any results provided for the study.

# 9. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Data is anonymized and extracted, analyzed, validated and reported in aggregate.

There is no potential that any employee of BI or agent working on behalf of BI will access individual patient data in which the patient may be identified during data compilation, data reporting or data analysis.

Based on current guidelines from the International Society for Pharmacoepidemiology [R11-4318] and the EMA [R13-1970], non-interventional studies such as the one described in this protocol, conducted using health care records, do not require expedited reporting of suspected adverse events/reactions. Specifically, as stated in section VI.C.1.2.1 of Guideline on Good Pharmacovigilance Practices (GVP), Module VI – Management and Reporting of Adverse Reactions to Medicinal Products, for non-interventional study designs, which are based on use of secondary data, reporting of adverse reactions is not required.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10. PLANS FOR DISSEMINATION AND COMMUNICATION OF STUDY RESULTS

We plan to publish the study in a peer-reviewed medical journal.

Authorship and publication will follow the corresponding BI SOP 001-MCS-00-002 and guidelines of good scientific practice.

#### 11. REFERENCES

#### 11.1 PUBLISHED REFERENCES

- P07-09514 Ernst P, Gonzalez AV, Brassard P, Suissa S. Inhaled corticosteroid use in chronic obstructive pulmonary disease and the risk of hospitalization for pneumonia. Am J Respir Crit Care Med 2007;176(2):162-166.
- P07-11503 Rabe KF, Hurd S, Anzueto A et al. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med 2007; 176(6):532-555.
- P14-12233 Kern DM, Williams SA, Tunceli O, Wessman C, Zhou S, Pethick N, Elhefni H, Trudo F. A US database study characterizing patients initiating a budesonide-fomoterol combination versus tiotropium bromide as initial maintenance therapy for chronic obstructive pulmonary disease. Int J COPD. 2014;(9): 775-783
- P14-13078 Rossi A, Guerriero M, Corrado A. Withdrawal of inhaled corticosteroids can be safe in COPD patients at low risk of exacerbation: a real-life study on the appropriateness of treatment in moderate COPD patients (OPTIMO). Respir Res 2014;15:77.
- P14-13477 Magnussen H, Disse B, Rodriguez-Roisin R et al. Withdrawal of inhaled glucocorticoids and exacerbations of COPD. N Engl J Med 2014;371(14):1285-1294.
- P15-08642 Barjaktarevic IZ, Arredondo AF, Cooper CB. Positioning new pharmacotherapies for COPD. Int J Chron Obstruct Pulmon Dis. 2015;10:1427-42. doi: 10.2147
- P15-11025 Trudo F, Kern DM, Davis JR. Comparative effectiveness of budesonide/formoterol combination and tiotropium bromide among COPD patients new to these controller treatments. Int J Chron Obstruct Pulmon Dis. 2015:10:2055–2066.
- P15-12888 Suissa S, Rossi A. Weaning from inhaled corticosteroids in COPD: the evidence. Eur Respir J 2015;46(5):1232-1235.
- P15-13167 Suissa S, Coulombe J, Ernst P. Discontinuation of Inhaled Corticosteroids in COPD and the Risk Reduction of Pneumonia. Chest 2015;148(5):1177-1183.
- P16-01440 Beeh KM, Derom E, Echave-Sustaeta J et al. The lung function profile of once-daily tiotropium and olodaterol via Respimat((R)) is superior to that of twice-daily salmeterol and fluticasone propionate via Accuhaler((R)) (ENERGITO((R)) study). Int J Chron Obstruct Pulmon Dis 2016;11:193-205.

- P16-05628 Wedzicha JA, Banerji D, Chapman KR et al. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med 2016;374(23):2222-2234.
- P16-10095 Suissa S, Dellaniello S, Ernst P. Long-acting bronchodilator initiation in COPD and the risk of adverse cardio-pulmonary events: A population-based comparative safety study. Chest 2017; 151(1):60-6
- P16-12287 Yawn BP, Suissa S, Rossi A. Appropriate use of inhaled corticosteroids in COPD: the candidates for safe withdrawal. NPJ Prim Care Respir Med 2016;26:16068.
- P17-04653 Suissa S, Moodie EE, Dell'Aniello S. Prevalent new-user cohort designs for comparative drug effect studies by time-conditional propensity scores. Pharmacoepidemiol Drug Saf 2017;26(4):459-468.
- P18-09975 Suissa S, Dell'Aniello S, Ernst P. Comparative effectiveness of LABA-ICS versus LAMA as initial treatment in COPD targeted by blood eosinophils: a population-based cohort study. Lancet Respir Med, 2018. 6(11): p. 855-862.
- R11-4318 Guidelines for Good Pharmacoepidemiology Practices (GPP) (revision 2: April 2007). http://www.pharmacoepi.org/resources/guidelines\_08027.cfm (access date: 13 September 2011); Bethesda: International Society for Pharmacoepidemiology (ISPE) (2007).
- R11-2162 Jick SS, Kaye JA, Vasilakis-Scaramozza C et al. Validity of the general practice research database. Pharmacotherapy 2003;23(5):686-689.
- R05-1384 Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017.
- R13-1383 Lopez AD, Shibuya K, Rao C et al. Chronic obstructive pulmonary disease: current burden and future projections. Eur Respir J 2006;27(2):397-412.
- European Medicines Agency (EMA), Heads of Medicines Agencies (HMA) Guideline on good pharmacovigilance practices (GVP): module VI management and reporting of adverse reactions to medicinal products (22 June 2012, EMA/873138/2011).
- R13-4036 Minino AM, Xu J, Kochanek KD. Deaths: Preliminary data for 2008. National Vital Statistics Reports NCHS 2010;59(2).
- Schneeweiss S, Rassen JA, Glynn RJ, Myers J, Daniel GW, Singer J, Solomon DH, Kim SJ, Rothman KJ, Liu J, Avorn J. Supplementing Claims Data with Outpatient Laboratory Test Results to Improve Confounding Adjustment in Effectiveness Studies of Lipid-Lowering Treatments. BMC Med Res Methodol. 2012;12:180.

- Quint JK, Mullerova H, DiSantostefano RL et al. Validation of chronic obstructive pulmonary disease recording in the Clinical Practice Research Datalink (CPRD-GOLD). BMJ Open 2014;4(7):e005540.
- R16-2198 Lawrenson R, Williams T, Farmer R. Clinical information for research; the use of general practice databases. J Public Health Med 1999;21(3):299-304.
- R18-2874 Lin J, Li Y, Tian H, Goodman MJ, Gabriel S, Nazareth T, et al. Costs and health care resource utilization among chronic obstructive pulmonary disease patients with newly acquired pneumonia.
- R19-2321 Stephenson JJ, Wertz D, Gu T, Patel J, Dalal AA. Clinical and economic burden of dyspnea and other chronic obstructive pulmonary disease symptoms in a managed care setting. Int J COPD, 2017; 12: 1947-1959.
- R19-2322 Ke X, Marvel J, Yu T-C, Wertz D, Geremakis C, Wang L, Stephenson JJ, Mannino DM. Impact of lung function on exacerbations, health care utilization, and costs among patients with COPD. Int J COPD, 2016; 11:1689-1703.
- R19-2323 Johannes CB, McQuay LJ, Midkiff KD, Calingaert B, Andrews EA, Tennis P, Brown JS, Camargo CA, Disantostefano R, Rothman KJ, Sturmer T, Lanes S, Davis KJ. The feasibility of using multiple databases to study rare outcomes: the potential effect of long-acting beta agonists with inhaled corticosteroid therapy on asthma mortality. Pharmacoepidemiology and Drug Safety 2017;26(4):446-458
- Wallace A, Kaila S, Bayer V, Shaikh A, Shinde MU, Willey V, Napier M, and Singer J. Health Care Resource Utilization and Exacerbation Rates in Patients with COPD Stratified by Disease Severity in a Commercially Insured Population. Journal of Managed Care & Specialty Pharmacy 2019 25:2, 205-217. Clinicoeconomics Outcomes Res. 2014; 6, 349 356.
- R19-3030 Desai, R.J., et al., A Propensity-score-based Fine Stratification Approach for Confounding Adjustment When Exposure Is Infrequent. Epidemiology, 2017. 28(2): p. 249-257.
- R19-3048 Miravitlles M, Anzueto A. Chronic Respiratory Infection in Patients with Chronic Obstructive Pulmonary Disease: What Is the Role of Antibiotics? Int J Mol Sci. 2017;18(7). pii: E1344. doi: 10.3390
- P19-08111 Calverley, P.M.A., et al., Triple Therapy in COPD: What We Know and What We Don't. COPD: Journal of Chronic Obstructive Pulmonary Disease, 2017. 14(6): p. 648-662.
- R19-3031 Lash, T.L., et al., Good practices for quantitative bias analysis. Int J Epidemiol, 2014. 43(6): p. 1969-85.

### Boehringer Ingelheim Protocol for non-interventional studies based on existing data

**BI Study Number 1237-0094** 

**** 

c30699487-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.2 UNPUBLISHED REFERENCES

None

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 12. FUNDING

There are no additional sources of funding.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 13. ANNEX

#### **ANNEX 1: LIST OF STAND-ALONE DOCUMENTS**

Documents listed in Annex 1 can be maintained separately from the study protocol. They should be clearly identifiable and provided on request. Write "None" if there is no document or list documents in a table as indicated below.

| Number | Document reference number | Date | Title |
|--------|---------------------------|------|-------|
| 1 | None | None | None |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2: ENCEPP CHECKLIST FOR STUDY PROTOCOLS

#### ENCePP Checklist for Study Protocols (Revision 2, amended)

Adopted by the ENCePP Steering Group on 14/01/2013

| Safety and effectiveness of maintenance treatment with Dlodaterol in comparison to maintenance treatment Corticosteroids, Long-acting β2 agonists and long-acting patients | with | a com | binatio | n of Inhale |
|---|---|---|---|---|
| Study reference number: 205.526 | | | | |
| Section 1: Milestones | Yes | No | N/A | <u>Page</u> |
| 1.1 Does the protocol specify timelines for 1.1.1 Start of data collection1 1.1.2 End of data collection2 1.1.3 Study progress report(s) 1.1.4 Interim progress report(s) 1.1.5 Registration in the EU PAS register 1.1.6 Final report of study results. | | | | Number(s) 15 15 15 15 15 |
| Comments: | | | | |
| Section 2: Research question | Yes | <u>No</u> | <u>N/A</u> | Page |
| 2.1Does the formulation of the research question and objectives clearly explain: 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) 2.1.2 The objective(s) of the study? 2.1.3 The target population? (i.e. population or subgroup to whom the study results are intended to be generalized) 2.1.4 Which formal hypothesis(-es) is (are) to be | | | | 17<br>17<br>17 |
| zvivi vimon ioinim njeomosis( os) is (mo) to oc | | | | |
| tested? 2.1.5 If applicable, that there is no a priori hypothesis? Comments: | | Ш | | |

<sup>1</sup> Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts. <sup>2</sup> Date from which the analytical dataset is completely available.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Section 3: Study design | | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 3.1 Is the study design described? (e.g. cohort, case-control, randomized controlled trial, new or alternative design) | | | | 18 |
| 3.2 Does the protocol specify the primary and secondary (if applicable) endpoint(s) to be investigated? | | | | 18 |
| 3.3 Does the protocol describe the measure(s) of effect? (e.g. relative risk, odds ratio, deaths per 1000 person-years, absolute risk, excess risk, incidence rate ratio, hazard ratio, number needed to harm (NNH) per year) | | | | 25-27 |
| Comments: | | | | |
| Section 4: Source and study populations | Yes | No | N/A | Page<br>Number(s) |
| 4.1Is the source population described? | | | | 18, 22 |
| 4.2Is the planned study population defined in terms of: 4.2.1 Study time period? 4.2.2 Age and sex? 4.2.3 Country of origin? 4.2.4 Disease/indication? 4.2.5 Co-morbidity? 4.2.6 Seasonality? | | | | 18<br>18<br>18<br>18, 22<br>18, 20-21<br>20 |
| 4.3 Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 18 |
| Comments: | | | | |
| Section 5: Exposure definition and measurement | | No | N/A | Page<br>Number(s) |
| 5.1 Does the protocol describe how exposure is defined and measured? (e.g. operational details for defining and categorizing exposure) | | | | 19 |
| 5.2 Does the protocol discuss the validity of exposure | | | | |

measurement? (e.g. precision, accuracy, prospective

ascertainment, exposure information recorded before

 $\boxtimes$ 

19, 22
# Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

c30699487-01

| Section 5: Exposure definition and measurement | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| the outcome occurred, use of validation sub-study) | | | | |
| 5.3 Is exposure classified according to time windows? (e.g. current user, former user, non-use) | $\boxtimes$ | | | 19 |
| 5.4 Is exposure classified based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | | |
| 5.5 Does the protocol specify whether a dose-<br>dependent or duration-dependent response is<br>measured? | | | | |
| Comments: | | | | |
| | _ | | | |
| Section 6: Endpoint definition and measurement | Yes | <u>No</u> | N/A | Page<br>Number(s) |
| 6.1 Does the protocol describe how the endpoints are defined and measured? | $\boxtimes$ | | | 19-20 |
| 6.2 Does the protocol discuss the validity of endpoint measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, prospective or retrospective ascertainment, use of validation substudy) | | | | 19-20, 22 |
| Comments: | | ı | | |
| Section 7: Confounders and effect modifiers | Yes | No | N/A | Page<br>Number(s) |
| <ul><li>7.1 Does the protocol address known confounders?</li><li>(e.g. collection of data on known confounders, methods of controlling for known confounders)</li></ul> | | | | 20-21 |
| 7.2 Does the protocol address known effect modifiers? (e.g. collection of data on known effect modifiers, anticipated direction of effect) | | | | 22 |
| Comments: | | | | |

| 8.1 Does the protocol describe the data source(s) used in the study for the ascertainment of: 8.1.1 Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, faceto-face interview, etc.) 8.1.2 Endpoints? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics, etc.) 8.1.3 Covariates? | |
|---|---|
| 8.1.1 Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, faceto-face interview, etc.) 8.1.2 Endpoints? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics, etc.) 8.1.3 Covariates? | |
| 8.1.2 Endpoints? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics, etc.) 8.1.3 Covariates? | |
| markers or values, claims data, self-report, patient interview including scales and questionnaires, vital statistics, etc.) 8.1.3 Covariates? | |
| 8.2 Does the protocol describe the information | |
| 8.2.1 Exposure? (e.g. date of dispensing, drug quantity, dose, number of days of supply | |
| prescription, daily dosage, prescriber) | |
| 8.2.2 Endpoints? (e.g. date of occurrence, multiple event, severity measures related to event) | |
| 8.2.3 Covariates? (e.g. age, sex, clinical and drug use history, co-morbidity, co-medications, life style, etc.) | |
| 8.3 Is a coding system described for: | |
| 8.3.1 Diseases? (e.g. International Classification of Diseases (ICD)-10) | |
| 8.3.2 Endpoints? (e.g. Medical Dictionary for | |
| Regulatory Activities (MedDRA) for adverse events) | |
| 8.3.3 Exposure? (e.g. WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC)Classification System) | |
| 8.4 Is the linkage method between data sources described? (e.g. based on a unique identifier or other) | |
| Comments: | _ |
| Section 9: Study size and power Yes No N/A Page Number(s) | |
| 9.1 Is sample size and/or statistical power calculated? | |
| Comments: | |

# Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

c30699487-01

| Section 10: Analysis plan | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 10.1 Does the plan include measurement of excess risks? | $\boxtimes$ | | | 25-27 |
| 10.2 Is the choice of statistical techniques described? | $\boxtimes$ | | | 25-27 |
| 10.3 Are descriptive analyses included? | $\boxtimes$ | | | 25 |
| 10.4 Are stratified analyses included? | $\boxtimes$ | | | 25-27 |
| 10.5 Does the plan describe methods for adjusting for confounding? | $\boxtimes$ | | | 25-27 |
| 10.6 Does the plan describe methods addressing effect modification? | $\boxtimes$ | | | 25-27 |
| Comments: | | | | |
| Section 11: Data management and quality control | Yes | No | N/A | Page<br>Number(s) |
| 11.1 Is information provided on the management of missing data? | | | | 22 |
| 11.2 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) | | | | 24 |
| 11.3 Are methods of quality assurance described? | $\boxtimes$ | | | 24 |
| 11.4 Does the protocol describe possible quality issues related to the data source(s)? | | | | 24 |
| 11.5 Is there a system in place for independent review of study results? | $\boxtimes$ | | | 27 |
| Comments: | | | | |
| Section 12: Limitations | Yes | No | N/A | Page<br>Number(s) |
| 12.1 Does the protocol discuss: 12.1.1 Selection biases? | | | $\boxtimes$ | |
| 12.1.2 Information biases? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods) | | | | 22, 28 |
| 12.2 Does the protocol discuss study feasibility? (e.g. sample size, anticipated exposure, duration of | $\boxtimes$ | | | 22-23 |

## Protocol for non-interventional studies based on existing data BI Study Number 1237-0094

c30699487-01

| Section 12: Limitations | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| follow-up in a cohort study, patient recruitment) | | | | |
| 12.3 Does the protocol address other limitations? | $\boxtimes$ | | | 22, 28 |
| Comments: | | | | |
| Section 13: Ethical issues | Yes | No | N/A | Page<br>Number(s) |
| 13.1 Have requirements of Ethics<br>Committee/Institutional Review Board approval been<br>described? | | | | 28-29 |
| 13.2 Has any outcome of an ethical review procedure been addressed? | | | | |
| 13.3 Have data protection requirements been described? | | | | 24 |
| Comments: | | | • | |
| Section 14: Amendments and deviations | Yes | No | N/A | Daga |
| Section 14. Amendments and deviations | 168 | 110 | IVIA | Page<br>Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? | | | | 14 |
| Comments: | | | | |
| C. d. 15. Diagram of the language | <b>X</b> 7 | NT - | NT/A | D |
| Section 15: Plans for communication of study results | Yes | No | N/A | Page<br>Number(s) |
| 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? | | | | |
| 15.2 Are plans described for disseminating study results externally, including publication? | | | | 29 |
| Comments: | | | | |
| Name of the main author of the protocol:<br>Date: 16 August 2019 | | | | |
| Signature: | | | | |

#### **ANNEX 3:ADDITIONAL INFORMATION**

Additional annexes may be included if necessary.

#### **ANNEX 3.1: DEFINITION OF STUDY EXPOSURES**

| Medication | HCPCS | GPI |
|---|---|---|
| LABA (single) | | |
| Indacaterol | | 44201042X |
| Salmeterol | | 4420105810X |
| Formoterol | J7605, J7606,<br>J7640, Q4099 | 44201027X 44201012102520 |
| Olodaterol | | 44201052X |
| LAMA (single) | | |
| Tiotropium | | 44100080X |
| Aclidinium | | 44100007X |
| Glycopyrronium | J7642, J7643 | 44100020X |
| Umeclidinium | | 44100090X |
| Revefenacin | | 44100075002020 |
| ICS (single) | | 4440X |
| | | 4220X |
| Fluticasone | J7641 | 44400033X |
| Budesonide | J7626, J7627,<br>J7633, J7634 | 44400015X |
| Beclomethasone | J7622 | 42200010x |
| | | 44400010x |
| Mometasone | | 42200045101820 |
| | | 44400036X |
| Flunisolide | J7641 | 44400030X |
| Ciclesonide | | 4440001700x |
| Dexamethasone | | 4440002010x |
| Triamcinolone | J7683, J7684 | 4440004020x |
| LABA/LAMA | | |
| Formoterol/glycopyrroni<br>um | | 44209902543220 |

| Medication | HCPCS | GPI |
|----------------------------------------------|-------|----------------|
| Indacaterol/glycopyrroni<br>um | | 44209902600110 |
| Vilanterol/umeclidinium | | 4420990295X |
| Olodaterol/tiotropium | | 4420990292X |
| LABA-LAMA-ICS | | |
| Fluticasone furoate/umeclidinium/vil anterol | | 44209903408020 |

### **ANNEX 3.2: DEFINITIONS OF STUDY OUTCOMES**

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10<br>proc | HCPCS | CPT |
|-----------|--------|--------|--------------|---------------|-------|-----|
| COPD | 491 | J41 | | | | |
| | 491 | J41.0 | | | | |
| | 491.1 | J41.1 | 1 | | | |
| | 491.2 | J41.8 | 1 | | | |
| | 491.21 | J42 | | | | |
| | 491.22 | J43 | | | | |
| | 491.8 | J43.0 | | | | |
| | 491.9 | J43.1 | | | | |
| | 492 | J43.2 | | | | |
| | 492 | J43.8 | | | | |
| | 492.8 | J43.9 | | | | |
| | 496 | J44 | | | | |
| | | J44.0 | | | | |
| | | J44.1 | | | | |
| | | J44.9 | | | | |
| Pneumonia | 480 | J10.00 | | | | |
| | 480.1 | J10.01 | | | | |
| | 480.2 | J10.08 | | | | |
| | 480.3 | J11.00 | | | | |

| 480.8 | J11.08<br>J12.0 |
|--------|-----------------|
| 481 | J12.1 |
| 482 | J12.2 |
| 482.1 | J12.3 |
| 482.2 | J12.81 |
| 482.3 | J12.89 |
| 482.31 | J12.9 |
| 482.32 | J13 |
| 482.39 | J14 |
| 482.4 | J15.0 |
| 482.41 | J15.3 |
| 482.42 | J15.4 |
| 482.49 | J15.5 |
| 482.81 | J15.6 |
| 482.82 | J15.7 |
| 482.83 | J15.8 |
| 482.84 | J15.9 |
| 482.89 | J16.0 |
| 482.9 | J16.8 |
| 483 | J17 |
| 483.1 | J18.0 |
| 483.8 | J18.1 |
| 484.1 | J18.2 |
| 484.3 | J18.8 |
| 484.5 | J18.9 |
| 484.6 | J69.0 |
| 484.7 | J85.1 |
| 484.8 | J95.4 |
| 485 | J95.89 |
| 486 | |
| 997.31 | |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

|--|

| Medication | HCPCS | GPI |
|--------------|---------------------|----------------|
| Prednisolone | J2650, J7510, J7512 | 22100040X |
| | | 22109902201810 |
| | | 22100045X |

#### **ANNEX 3.3: DEFINITIONS OF STUDY COVARIATES**

Complete list of ICD-9-CM, ICD-10, CPT, HCPCS, and GPI codes.

| Medication | HCPCS | GPI |
|---|---|---|
| Short-acting beta-<br>agonists | | |
| Levalbuterol | J7617,J7607,J7612, | 4420104510X |
| | J7614,J7615 | 4420104550X |
| Albuterol | J7602, J7603, | 4420101000X |
| | J7609-J7611, | 4420101010X |
| | J7613, J7616,<br>J7620, | |
| | J7625, Q4093,<br>Q4094 | |
| Terbutaline | J3105,J7680,J7681 | 442010602X |
| Isoproterenol | J7657 | 44201040X |
| | J7658 | |
| | J7659 | |
| | J7660 | |
| Methylxanthines | | |
| Aminophylline | | 4430001000x |
| | | 4430001010x |
| Theophylline (SR) | J2810 | 4430004000x 499100240X |
| | | 4499100220X |
| | | 4499100242X 4499100250X<br>44992203X |
| | | 44993003X 44993204X 44999003X |
| | | 44999602X 4499220310X |
| | | 4499960270X |
| | | 4499220315X |

| Medication | HCPCS | GPI |
|--------------------------------------------|--------------|-----------------|
| SAMA (Short-acting muscarinic antagonists) | | |
| Ipratropium bromide | J7644, J7655 | 4230X 44100030X |
| Antibiotics for a respiratory condition | | |
| Aamikacin | J0278 | 07000010x |
| Amoxicillin/potassium clavulanate | | 0199000220x |
| Amoxicillin | | 01200010x |
| Ampicillin | J0290 | 01200020x |
| Ampicillin-sulbactam | J0295 | 0199000225x |
| Azithromycin | J0456 | 03400010x |
| Aztreonam | S0073 | 16000005x |
| Cefaclor | | 02200040x |
| Cefdinir | | 02300040x |
| Cefepime | J0692 | 02400040x |
| Cefixime | | 02300060x |
| Cefotaxime | J0698 | 02300075x |
| Cefpodoxime | | 02300065x |
| Cefprozil | | 02200062x |
| Ceftazidime | J0713, J0714 | 02300080x |
| Ceftriaxone | J0696 | 02300090x |
| Cefuroxime | J0697 | 02200065x |
| Ciprofloxacin | J0744 | 05000020x |
| Clarithromycin | | 03500010x |
| Doxycycline | | 04000020x |
| Ertapenem | J1335 | 16150030x |
| Erythromycin | J1364 | 0310x |
| Gemifloxacin | | 05000083x |
| Imipenem | J0743 | 16159902x |
| Levofloxacin | J1956 | 05000034x |
| Linezolid | J2020 | 16230040x |

| Medication | HCPCS | GPI |
|-----------------------------------|--------------|----------------------|
| Meropenem | J2185 | 16150050x |
| Moxifloxacin | J2280 | 05000037x |
| Penicillin G benzathine | J0561, J0558 | 01990002x, 01100020x |
| Penicillin VK | | 01100040x |
| Piperacillin | S0081 | 01400040x |
| Piperacillin-tazobactam | J2543 | 019900027x |
| Procaine penicillin | J0558, J2510 | |
| Ticarcillin | | 01400050x |
| Ticarcillin-clavulanate | S0040 | 019900023x |
| Trimethoprim-<br>sulfamethoxazole | S0039 | 169900023x |
| Vancomycin | J3370 | 16000060102x |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|-----------|--------|--------|--------------|------------|-----------|-----|
| Asthma | 493 | J45 | | | | |
| | 493 | J45.2 | | | | |
| | 493 | J45.20 | | | | |
| | 493.01 | J45.21 | | | | |
| | 493.02 | J45.22 | | | | |
| | 493.1 | J45.3 | | | | |
| | 493.1 | J45.30 | | | | |
| | 493.11 | J45.31 | | | | |
| | 493.12 | J45.32 | | | | |
| | 493.2 | J45.4 | | | | |
| | 493.2 | J45.40 | | | | |
| | 493.21 | J45.41 | | | | |
| | 493.22 | J45.42 | | | | |
| | 493.8 | J45.5 | | | | |
| | 493.81 | J45.50 | | | | |
| | 493.82 | J45.51 | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | 493.9 | J45.52 | | | | |
| | 493.9 | J45.9 | | | | |
| | 493.91 | J45.90 | | | | |
| | 493.92 | J45.901 | | | | |
| | | J45.902 | 1 | | | |
| | | J45.909 | 1 | | | |
| | | J45.99 | 1 | | | |
| | | J45.990 | | | | |
| | | J45.991 | 1 | | | |
| | | J45.998 | | | | |
| Interstitial lung disease | 162<br>231.2<br>197.0<br>176.4<br>235.7<br>V10.11<br>516.6*<br>516.34 | C33 C34.00 C34.10 C34.2 C34.30 C34.80 C34.90 C46.50 C78.00 D02.20 D38.1 Z85.118 J84.115 J84.83 J84.841 | | | | |
| Lung | | J84.842<br>J84.843<br>J84.848 | 33.50 | 0BYC0Z0 | S2060 | 00580 |
| transplant | | | 33.51 | 0BYC0Z1 | S2061 | 32850 |
| | | | 33.52 | 0BYC0Z2 | | 32856 |
| | | | | 0BYD0Z0 | | 33935 |
| | | | | 0BYD0Z1 | - | 33933 |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | | | | 0BYD0Z2 | | |
| | | | | 0BYF0Z0 | 1 | |
| | | | | 0BYF0Z1 | 1 | |
| | | | | 0BYF0Z2 | | |
| | | | | 0BYG0Z0 | | |
| | | | | 0BYG0Z1 | | |
| | | | | 0BYG0Z2 | | |
| | | | | 0BYH0Z0 | | |
| | | | | 0BYH0Z1 | | |
| | | | | 0BYH0Z2 | | |
| | | | | 0BYJ0Z0 | | |
| | | | | 0BYJ0Z1 | | |
| | | | | 0BYJ0Z2 | | |
| | | | | 0BYK0Z0 | | |
| | | | | 0BYK0Z1 | | |
| | | | | 0BYK0Z2 | | |
| | | | | 0BYL0Z0 | | |
| | | | | 0BYL0Z1 | | |
| | | | | 0BYL0Z2 | | |
| | | | | 0BYM0Z0 | | |
| | | | | 0BYM0Z1 | | |
| | | | | 0BYM0Z2 | | |
| Cardiovascul<br>ar disease | 410.xx-<br>414.xx<br>427.xx;<br>785.0; 785.1<br>426.xx<br>428.xx<br>401.xx-<br>405.xx<br>440.xx;<br>441.xx;<br>442.xx; | 120.%-<br>125.%%%<br>147.%,<br>148.%%;<br>149.%%<br>144.%%;<br>145.%%<br>150.%%<br>111.%;<br>113.%;<br>O10.1%;<br>O10.3% | 37.7x-<br>37.8x,<br>37.94-<br>37.99 | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | 443.xx<br>272.x<br>393-398;<br>421.x;<br>422.xx;<br>746.0x-746.7 | I70.%%%;<br>I71.%%;<br>I72.%;<br>I73.%%<br>E78.%%<br>I05.%-<br>I09.%%;<br>I33.%-I39;<br>Q22.%,<br>Q23.% | 1 | | | |
| Diabetes | 250 | E10.10 | | | | |
| | 250.01 | E10.11 | | | | |
| | 250.02 | E10.21 | | | | |
| | 250.03 | E10.29 | | | | |
| | 250.1 | E10.311 | | | | |
| | 250.11 | E10.319 | | | | |
| | 250.12 | E10.36 | | | | |
| | 250.13 | E10.37X1 | | | | |
| | 250.2 | E10.37X2 | | | | |
| | 250.21 | E10.37X3 | | | | |
| | 250.22 | E10.37X9 | | | | |
| | 250.23 | E10.39 | | | | |
| | 250.3 | E10.40 | | | | |
| | 250.31 | E10.51 | | | | |
| | 250.32 | E10.618 | | | | |
| | 250.33 | E10.620 | | | | |
| | 250.4 | E10.621 | ] | | | |
| | 250.41 | E10.622 | ] | | | |
| | 250.42 | E10.628 | | | | |
| | 250.43 | E10.630 | | | | |
| | 250.5 | E10.638 | | | | |
| | 250.51 | E10.641 | | | | |
| | 250.52 | E10.649 | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | 250.53 | E10.65 | | | | |
| | 250.6 | E10.69 | | | | |
| | 250.61 | E10.10 | | | | |
| | 250.62 | E10.11 | | | | |
| | 250.63 | E10.21 | | | | |
| | 250.7 | E10.29 | | | | |
| | 250.71 | E10.311 | | | | |
| | 250.72 | E10.319 | | | | |
| | 250.73 | E10.36 | | | | |
| | 250.8 | E10.37X1 | | | | |
| | 250.81 | E10.37X2 | | | | |
| | 250.82 | E10.37X3 | | | | |
| | 250.83 | E10.37X9 | | | | |
| | 250.9 | E10.39 | | | | |
| | 250.91 | E10.40 | | | | |
| | 250.92 | E10.51 | | | | |
| | 250.93 | E10.618 | | | | |
| | | E10.620 | | | | |
| | | E10.621 | | | | |
| | | E10.622 | | | | |
| | | E10.628 | | | | |
| | | E10.630 | | | | |
| | | E10.638 | | | | |
| | | E10.641 | | | | |
| | | E10.649 | | | | |
| | | E10.65 | | | | |
| | | E10.69 | | | | |
| | | E10.10 | | | | |
| | | E10.11 | | | | |
| | | E10.21 | | | | |
| Thyroid | 226, 240.0, | D09.3, D34, | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | CPT |
|---|---|---|---|---|---|---|
| disease | 240.9, 241.0,<br>241.1, 241.9,<br>242*, 243,<br>244*, 245*,<br>246*, 790.94 | D44.0,<br>E01.1,E01.2,<br>E01.8, E02,<br>E03*, E04*,<br>E05*, E06*,<br>E07*,<br>E01.0<br>E89.0 | | | | |
| Renal failure | 403 | I12.0 | | | | |
| | 403.01 | I12.9 | | | | |
| | 403.1 | N18.1 | | | | |
| | 403.11 | N18.2 | | | | |
| | 403.9 | N18.3 | | | | |
| | 403.91 | N18.4 | | | | |
| | 585.1 | N18.5 | | | | |
| | 585.2 | N18.6 | | | | |
| | 585.3 | N18.9 | | | | |
| | 585.4 | N17.0 | | | | |
| | 585.5 | N17.1 | | | | |
| | 585.6 | N17.2 | | | | |
| | 585.9 | N17.8 | | | | |
| | 586 | N17.9 | | | | |
| Autoimmune | 135 | D86.9 | | | | |
| disease | 274.9 | M10.9 | | | | |
| | 275.49 | E83.59 | | | | |
| | 279.49 | D89.89 | | | | |
| | 283 | D59.0 | | | | |
| | 443 | D59.1 | | | | |
| | 448.9 | I73.00 | | | | |
| | 530.5 | I73.01 | | | | |
| | 555.9 | I78.9 | | | | |
| | 571.42 | K22.4 | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|-----------|--------|--------|--------------|------------|-----------|-----|
| | 571.6 | K50.90 | | | | |
| | 576.1 | K75.4 | | | | |
| | 579 | K74.3 | | | | |
| | 696 | K74.4 | | | | |
| | 696.1 | K74.5 | | | | |
| | 710 | K83.0 | | | | |
| | 710.1 | K90.0 | | | | |
| | 710.2 | L40.50 | | | | |
| | 710.3 | L40.54 | | | | |
| | 710.9 | L40.59 | | | | |
| | 711.9 | L40.0 | | | | |
| | 712.19 | L40.1 | | | | |
| | 714 | L40.2 | | | | |
| | 714.3 | L40.8 | | | | |
| | 715.09 | M32.10 | | | | |
| | 715.11 | M34.0 | | | | |
| | 715.12 | M34.1 | | | | |
| | 715.13 | M34.2 | | | | |
| | 715.14 | M34.81 | | | | |
| | 715.15 | M34.82 | | | | |
| | 715.17 | M34.83 | | | | |
| | 715.18 | M34.89 | | | | |
| | 715.96 | M34.9 | | | | |
| | 719.42 | M35.00 | | | | |
| | 719.44 | M35.01 | | | | |
| | 719.45 | M35.02 | | | | |
| | 719.47 | M35.03 | | | | |
| | 719.49 | M35.04 | | | | |
| | 720 | M35.09 | | | | |
| | 721.9 | M33.90 | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | CPT |
|-----------|--------|---------|--------------|------------|-----------|-----|
| | 725 | M35.9 | | | | |
| | 729.1 | M00.9 | | | | |
| | 729.5 | M11.9 | | | | |
| | 795.79 | M06.9 | | | | |
| | | M08.00 | | | | |
| | | M15.0 | | | | |
| | | M19.019 | | | | |
| | | M19.029 | | | | |
| | | M19.039 | | | | |
| | | M19.049 | | | | |
| | | M16.0 | | | | |
| | | M16.10 | | | | |
| | | M16.11 | | | | |
| | | M16.12 | | | | |
| | | M19.079 | | | | |
| | | M19.91 | | | | |
| | | M17.9 | | | | |
| | | M25.529 | | | | |
| | | M79.643 | | | | |
| | | M79.646 | | | | |
| | | M25.559 | | | | |
| | | M25.579 | | | | |
| | | M25.50 | | | | |
| | | M45.9 | | | | |
| | | M47.819 | | | | |
| | | M35.3 | | | | |
| | | M60.9 | | | | |
| | | M79.1 | ] | | | |
| | | M79.609 | ] | | | |
| | | R76.0 | | | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | | R76.11 | | | | |
| | | R76.12 | | | | |
| | | R76.8 | | | | |
| | | R76.9 | | | | |
| Obesity | 278 | E65 | | | | |
| | 278.01 | E66.01 | | | | |
| | 278.02 | E66.2 | | | | |
| | 278.03 | E66.3 | | | | |
| | 278.1 | E66.9 | | | | |
| | 278.2 | E67.0 | | | | |
| | 278.3 | E67.1 | | | | |
| | 278.4 | E67.3 | | | | |
| | 278.8 | E67.8 | | | | |
| | V85.30 | Z68.30 | | | | |
| | V85.31 | Z68.31 | | | | |
| | V85.32 | Z68.32 | | | | |
| | V85.33 | Z68.33 | | | | |
| | V85.34 | Z68.34 | | | | |
| | V85.35 | Z68.35 | | | | |
| | V85.36 | Z68.36 | | | | |
| | V85.37 | Z68.37 | | | | |
| | V85.38 | Z68.38 | | | | |
| | V85.39 | Z68.39 | | | | |
| Alcohol use disorder | 303 | F10.159 | 94.46 | HZ2ZZZ<br>Z | | |
| | 303.01 | F10.180 | 94.53 | HZ30ZZ<br>Z | | |
| | 303.02 | F10.181 | 94.61 | HZ31ZZ<br>Z | | |
| | 303.03 | F10.188 | 94.62 | HZ32ZZ<br>Z | | |
| | 303.9 | F10.20 | 94.63 | HZ33ZZ | | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|-----------|--------|---------|--------------|-------------|-----------|-----|
| | | | | Z | | |
| | 303.91 | F10.21 | 94.67 | HZ34ZZ<br>Z | | |
| | 303.92 | F10.229 | 94.68 | HZ35ZZ<br>Z | | |
| | 303.93 | F10.259 | 94.69 | HZ36ZZ<br>Z | | |
| | | F10.27 | | HZ37ZZ<br>Z | | |
| | | F10.280 | | HZ38ZZ<br>Z | | |
| | | F10.281 | | HZ39ZZ<br>Z | | |
| | | F10.288 | | HZ3BZZ<br>Z | | |
| | | F10.959 | | HZ40ZZ<br>Z | | |
| | | F10.980 | | HZ41ZZ<br>Z | | |
| | | F10.99 | | HZ42ZZ<br>Z | | |
| | | Z65.8 | | HZ43ZZ<br>Z | | |
| | | | | HZ44ZZ<br>Z | - | |
| | | | | HZ45ZZ<br>Z | - | |
| | | | | HZ46ZZ<br>Z | | |
| | | | | HZ47ZZ<br>Z | | |
| | | | | HZ48ZZ<br>Z | | |
| | | | | HZ49ZZ<br>Z | | |
| | | | | HZ4BZZ<br>Z | - | |

| Condition | ICD9 | ICD10 | ICD9<br>proc | ICD10 proc | HCPC<br>S | СРТ |
|---|---|---|---|---|---|---|
| | | | | HZ93ZZ<br>Z | | |
| | | | | HZ96ZZ<br>Z | | |
| Tobacco use or cessation counselling | 305.1*<br>649.0*<br>989.84<br>V15.82 | Z72.0<br>F17.21<br>F17.210<br>F17.211<br>F17.218<br>F17.219<br>Z71.6 | | | C9801<br>C9802<br>G0375<br>G0376<br>G0436<br>G0437<br>G8453<br>G8455<br>G8456<br>G8692<br>G9276<br>G9458<br>G9497<br>G9642<br>G9792<br>G9906<br>G9908<br>S9075<br>S9453<br>G9902<br>G9907<br>G9909 | 99406 99407 |
| Cancer (excluding basal cell | 140.xx -<br>195.xx | C00%-C76%, | | | | |
| carcinoma) | 200.xx –<br>208.xx | C81%-C96% | | | | |
| | 196.xx -<br>199.xx | C77%-C80% | | | | |
| | EXCLUDIN<br>G: | EXCLUDIN<br>G: | | | | |
| | 173.01 | C44.01 | | | | |
| | 173.11 | C44.111 | | | | |

| Condition | ICD9 | ICD10 | ICD9 | ICD10 proc | HCPC | CPT |
|-----------|--------|----------|------|------------|------|-----|
| | | | proc | | S | |
| | 173.21 | C44.1121 | | | | |
| | 173.31 | C44.119 | | | | |
| | 173.41 | C44.91 | | | | |
| | 173.51 | C44.311 | | | | |
| | 173.61 | C44.319 | | | | |
| | 173.71 | C44.310 | | | | |
| | 173.81 | C44.510 | | | | |
| | 173.91 | C44.511 | | | | |
| | | C44.519 | | | | |
| | | C44.41 | | | | |
| | | C44.81 | | | | |
| | | C44.211 | | | | |
| | | C44.212 | | | | |
| | | C44.219 | | | | |
| | | C44.611 | | | | |
| | | C44.612 | | | | |
| | | C44.619 | | | | |
| | | C44.711 | | | | |
| | | C44.712 | | | | |
| | | C44.719 | | | | |

### **ANNEX 3.4:STATISTICAL CONSIDERATIONS**

See section 7.9



#### APPROVAL / SIGNATURE PAGE

Document Number: c30699487 Technical Version Number: 1.0

Document Name: bi-se-laba-tt-final

**Title:** Effectiveness and Safety of Maintenance Treatment with Combination of Tiotropium and Olodaterol in comparison to Maintenance Treatment with a Combination of Inhaled Corticosteroids, Long-acting β2 Agonists and Long-acting Muscarinic Antagonists in COPD Patients

#### **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval-Other | | 17 Dec 2019 13:14 CET |
| Approval- Safety Evaluation<br>Therapeutic Area | | 18 Dec 2019 08:50 CET |
| Approval- of Global<br>Epidemiology | | 07 Jan 2020 20:03 CET |
| Approval-Team Member Medicine | | 16 Jan 2020 14:11 CET |
| Approval-Team Member Medicine | | 16 Jan 2020 15:26 CET |

Boehringer IngelheimPage 2 of 2Document Number: c30699487Technical Version Number:1.0

### (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|